CLINICAL TRIAL: NCT00770471
Title: A Phase I/II Trial of Temozolomide and ABT-888 in Subjects With Newly Diagnosed Glioblastoma Multiforme
Brief Title: ABT-888, Radiation Therapy, and Temozolomide in Treating Patients With Newly Diagnosed Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NABTT-0801 CDR0000616542; U01CA062475 (NIH); ABTC-0801; NABTT-0801; ABBOTT-M10-190
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult gliosarcoma; adult giant cell glioblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — Temozolomide; veliparib; DNA Methylation; Gene Expression Profiling; Chromatography, High Pressure Liquid; Immunoenzyme Techniques; Mass Spectrometry; Pharmacogenomic Testing; Chemotherapy, Adjuvant; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental)
  Interventions: Drug: temozolomide; Drug: veliparib; Genetic: DNA methylation analysis; Genetic: gene expression analysis; Genetic: mutation analysis; Genetic: proteomic profiling; Other: high performance liquid chromatography; Other: immunoenzyme technique; Other: laboratory biomarker analysis; Other: mass spectrometry; Other: pharmacogenomic studies; Other: pharmacological study; Procedure: adjuvant therapy; Radiation: radiation therapy

INTERVENTIONS:
Drug: temozolomide
Drug: veliparib
Genetic: DNA methylation analysis
Genetic: gene expression analysis
Genetic: mutation analysis
Genetic: proteomic profiling
Other: high performance liquid chromatography
Other: immunoenzyme technique
Other: laboratory biomarker analysis
Other: mass spectrometry
Other: pharmacogenomic studies
Other: pharmacological study
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: ABT-888 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving ABT-888 together with radiation therapy and temozolomide may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of ABT-888 when given together with radiation therapy and temozolomide and to see how well it works in treating patients with newly diagnosed glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose (MTD) of ABT-888 when administered in combination with radiotherapy and temozolomide in patients with newly diagnosed glioblastoma multiforme. (Phase I)
* To estimate the overall survival of patients treated with ABT-888 when administered at the MTD in combination with radiotherapy and temozolomide. (Phase II)

Secondary

* To assess the toxicity associated with this regimen. (Phase I)
* To assess and describe the pharmacokinetics of ABT-888. (Phase I)
* To estimate the frequency of toxicity associated with this regimen. (Phase II)

OUTLINE: This is a multicenter, phase I dose-escalation study of ABT-888 followed by a phase II study.

* Initiation therapy: Patients receive oral ABT-888 twice daily (once on day 1 only) and oral temozolomide once daily (beginning on day 2) in weeks 1-6. Patients enrolled in the phase I dose-escalation/phase II portion of the study also undergo concurrent radiotherapy once daily 5 days a week (beginning on day 2) in weeks 1-6. Treatment continues in the absence of disease progression or unacceptable toxicity.
* Maintenance therapy: Beginning 4 weeks after completion of initiation therapy, patients receive oral ABT-888 twice daily on days 1-7 and oral temozolomide once daily on days 1-5. Treatment repeats every 28 days for up to 4 courses (6 courses for patients enrolled in the phase I dose-escalation/phase II portion of the study) in the absence of disease progression or unacceptable toxicity.

Blood samples are collected periodically for pharmacokinetic, pharmacogenetic, and pharmacodynamic analysis. Samples are analyzed for concentration of ABT-888 in plasma by reversed-phase isocratic high performance liquid chromatography with electrospray ionization mass spectrometry; identification of novel markers of treatment response by plasma proteomic evaluation; DNA methylation and/or mutation; and PARP inhibition by ELISA.

After completion of study therapy, patients are followed every 2 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed supratentorial grade IV astrocytoma (glioblastoma multiforme)

  * Newly diagnosed disease
* Patients enrolled in the phase I initial safety portion of the study must meet the following additional criteria:

  * Received 90% of planned radiotherapy and ≥ 80% of planned concurrent temozolomide within the past 28-49 days

    * No grade 3-4 toxicity attributed to temozolomide
  * Has undergone gadolinium MRI or contrast CT scan within the past 28 days
* Patients enrolled in the phase I dose-escalation/phase II portion of the study must meet the following additional criteria:

  * Recovered from immediate post-operative period and maintained on a stable corticosteroid regimen (no increase in 5 days) prior to starting study treatment
  * Has undergone gadolinium MRI or contrast CT scan within the past 14 days

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Life expectancy ≥ 3 months
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL
* Creatinine ≤ 2.0 mg/dL OR creatinine clearance ≥ 60 mL/min
* Total bilirubin ≤ 1.5 mg/dL
* Transaminases ≤ 2.5 times upper limit of normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception prior to, during, and for 3 months after completion of study therapy
* Mini Mental State Exam score ≥ 15
* Able to swallow and retain oral medications
* No concurrent serious infection or medical illness that would jeopardize the ability of the patient to receive study treatment with reasonable safety
* No other malignancy within the past 5 years except for curatively treated carcinoma in situ or basal cell carcinoma of the skin
* No known uncontrolled seizure disorder (i.e., status epilepticus) or seizures occurring ≥ 3 times per week over the past month

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 10 days since prior cytochrome P450-inducing anticonvulsants (e.g., phenytoin, carbamazepine, phenobarbital, primidone, or oxcarbazepine)
* At least 1 week since prior biopsy or resection of tumor (for patients enrolled in the phase I dose-escalation/phase II portion of the study)
* No prior radiotherapy, chemotherapy, immunotherapy, hormonal therapy, or biological therapy (including immunotoxins, immunoconjugates, antisense therapy, peptide receptor antagonists, interferons, interleukins, tumor-infiltrating lymphocytes, lymphokine-activated killer cells, or gene therapy) for treatment of brain tumor (for patients enrolled in the phase I dose-escalation/phase II portion of the study)

  * Prior glucocorticoid therapy allowed
* No other prior chemotherapy or investigational agents (for patients enrolled in the phase I initial safety portion of the study)
* Prior Gliadel wafers allowed (for patients enrolled in the phase I portion of the study)
* No prior Gliadel wafers (for patients enrolled in the phase II portion of the study)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-07-13 (Actual); Primary Completion 2012-03-01 (Actual); Study Completion 2012-03-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of ABT-888 (Phase I) | continous
Overall survival (Phase II) | continous

SECONDARY OUTCOMES:
Toxicity (Phase I) | continous
Pharmacokinetics of ABT-888 (Phase I) | continous
Frequency of toxicity (Phase II) | continous

CONTACTS AND LOCATIONS:
Overall Officials: Larry Kleinberg, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (11):
- United States (11):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No